CLINICAL TRIAL: NCT06789328
Title: The Effect of Dexamethasone Administration Route on Pain and Inflammatory Response in PENG Block for Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2/2025
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Hip; Hip Pain Chronic; Hip Arthropathy; Hip Arthritis
Keywords: pericapsular nerve group block; PENG block; adjuvant; dexamethasone
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perineural dexamethasone (Active Comparator): PENG block + perineural dexamethasone
  Interventions: Drug: perineural Dexamethasone 4mg
- Intravenous dexamethasone (Active Comparator): PENG block + intravenous dexamethasone
  Interventions: Drug: intravenous Dexamethsone 4mg

INTERVENTIONS:
Drug: perineural Dexamethasone 4mg — PENG block with 20ml 0.2% ropivacaine + 4mg perineural Dexamethasone
  Arms: Perineural dexamethasone
Drug: intravenous Dexamethsone 4mg — PENG block with 20ml 0.2% ropivacaine + 4mg intravenous Dexamethasone
  Arms: Intravenous dexamethasone

SUMMARY:
This study aims to evaluate the effect of the dexamethasone administration route (intravenous vs. perineural) on postoperative pain, inflammatory response, and clinical outcomes in patients undergoing total hip arthroplasty (THA) with a pericapsular nerve group (PENG) block. The primary outcome is the intensity of postoperative pain measured using the numerical rating scale (NRS) at rest and during movement. Secondary outcomes include the inflammatory response assessed by neutrophil-to-lymphocyte ratio (NLR) and platelet-to-lymphocyte ratio (PLR), opioid consumption, and patient satisfaction. The findings from this study may contribute to optimizing anesthesia protocols and improving postoperative recovery in patients undergoing THA.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a common orthopedic procedure associated with significant postoperative pain and inflammation, which can impact recovery and long-term outcomes. Regional anesthesia techniques, such as the pericapsular nerve group (PENG) block, have become increasingly popular for pain management in THA due to their ability to provide effective analgesia while preserving motor function.

Dexamethasone is frequently used as an adjuvant in regional anesthesia to prolong the duration of analgesia and reduce inflammation. However, there is limited evidence comparing the efficacy of different administration routes of dexamethasone (intravenous vs. perineural) in the context of PENG block. Additionally, understanding the impact of dexamethasone on postoperative pain, inflammatory markers, and overall patient recovery is crucial for optimizing clinical protocols.

This study is a prospective, randomized, double-blinded trial involving patients undergoing elective THA. Participants will be randomly assigned to two groups: the IV dexamethasone group or the perineural dexamethasone group. Both groups will receive standardized general anesthesia and PENG block with local anesthetic. Postoperative pain will be assessed using the NRS at various time intervals (e.g., 6, 12, 24, and 48 hours postoperatively) at rest and during movement. NLR and PLR will measure the inflammatory response from blood samples taken preoperatively and 24 hours postoperatively.

The primary outcome is time first to request rescue analgesia. Secondary outcomes include cumulative opioid consumption, length of hospital stay, and patient satisfaction. Safety and potential complications, such as local anesthetic systemic toxicity (LAST), will be closely monitored.

The results of this study may provide valuable insights into the optimal use of dexamethasone as an adjuvant in regional anesthesia for THA, potentially improving pain management, reducing opioid use, and enhancing postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total hip arthroplasty
* patients aged >65 and <100 years
* patients able to provide informed consent
* patients able to reliably report symptoms to the research team

Exclusion Criteria:

* inability to provide first-party consent due to cognitive impairment or a language barrier
* infection at the site of the regional block,
* coagulation disorders,
* immunodeficiency,
* American Society of Anesthesiologists (ASA) physical status of IV or higher,
* history of regular steroid medication.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Time to first rescue opioid analgesia | 48 hours after surgery
  Time to first rescue opioid analgesia

SECONDARY OUTCOMES:
Total opioid consumption | 48 hours after surgery
  Total opioid consumption (mg) converted to morphine milligram equivalents (MME)
NRS | 4 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NRS | 8 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NRS | 12 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NRS | 24 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NRS | 48 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NLR | 12 hours after surgery
  Neutrophil-to-lymphocyte ratio
NLR | 24 hours after surgery
  Neutrophil-to-lymphocyte ratio
NLR | 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 12 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 24 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 48 hours after surgery
  Platelet-to-lymphocyte ratio
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 4 hours after surgery
  uadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale.
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 8 hours after surgery
  uadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale.
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 12 hours after surgery
  uadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale.
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 24 hours after surgery
  uadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale.
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 48 hours after surgery
  uadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale.
Nerve damage | 12 hours after surgery
  Nerve damage assessment will be performed using the following grading scale:
  N0 - No nerve damage N1 - Minor: sensory paresthesia N2 - Major: complete sensory anesthesia N3 - Complete: complete motor deficit with or without paresthesia N4 - CRPS: Complex Regional Pain Syndrome
Nerve damage | 24 hours after surgery
  Nerve damage assessment will be performed using the following grading scale:
  N0 - No nerve damage N1 - Minor: sensory paresthesia N2 - Major: complete sensory anesthesia N3 - Complete: complete motor deficit with or without paresthesia N4 - CRPS: Complex Regional Pain Syndrome
Nerve damage | 48 hours after surgery
  Nerve damage assessment will be performed using the following grading scale:
  N0 - No nerve damage N1 - Minor: sensory paresthesia N2 - Major: complete sensory anesthesia N3 - Complete: complete motor deficit with or without paresthesia N4 - CRPS: Complex Regional Pain Syndrome
glucose | 12 hours after surgery
  blood glucose level
glucose | 24 hours after surgery
  blood glucose level
glucose | 48 hours after surgery
  blood glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, M.D. Ph.D., Study Chair — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland